CLINICAL TRIAL: NCT05058469
Title: Evaluation of the Safety of Percutaneous Tracheotomies in Intensive Care Patients With and Without Antiplatelet Therapy and Comparison of Two Tracheotomy Techniques
Brief Title: Tracheotomy With and Without Dual Antiplatelet Therapy
Acronym: PDT and (D)APT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asklepios Neurological Clinic Bad Salzhausen (Other)
Responsible Party: Sponsor
Other Study IDs: PDT and (D)APT
Record Dates: First submitted 2021-09-14; First posted 2021-09-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-12

CONDITIONS: Tracheostomy Hemorrhage
MeSH Terms: interventions — Tracheotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Tracheotomy without antiplatelet therapy+technique 1
  Interventions: Device: Tracheotomy
- Tracheotomy under antiplatelet therapy+technique 1
  Interventions: Device: Tracheotomy
- Tracheotomy without antiplatelet therapy+technique 2
  Interventions: Device: Tracheotomy
- Tracheotomy under antiplatelet therapy+technique 2
  Interventions: Device: Tracheotomy

INTERVENTIONS:
Device: Tracheotomy — Tracheotomy in patients +/- antiplatelet therapy

SUMMARY:
Platelet-inhibiting drugs are often used after vascular interventions. Patients who require such therapies are often critically ill, are treated in intensive care units and often require long-term ventilation. For long-term ventilation a tracheotomy is necessary, which is usually performed as a percutaneous dilatative tracheotomy (PDT). As part of this intervention, there is (theoretically) an increased risk of bleeding/an increased rate of complications in patients with a antiplatelet therapy. In addition, there are various techniques for performing a PDT.

The current study aims to investigate the frequency of bleeding/complications taking into account the technique used in PDT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Percutaneous Dilational Tracheostomy

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent Percutaneous Dilational Tracheostomy within the last 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of bleeding during Percutaneous Dilational Tracheostomy (PDT) with and without antiplatelet therapy (AP). | 3 days
  * bleeding (yes/no)
  * intervention (yes/no)
  * decrease (>= 1 g/dl) of hemoglobin (yes/no)
  * number of blood transfusion(s)

SECONDARY OUTCOMES:
- Does the technique of PDT affect the bleeding rate? - How often are recognizable cartilage pin fractures in the context of a PDT? - Influence of AP and PDT technology on the frequency of need for a blood transfusion? | 14 days
  cartilage pin fractures seen in endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Neurologische Klinik Bad Salzhausen, Nidda, Germany

IPD SHARING:
Plan to Share IPD: No